CLINICAL TRIAL: NCT05028504
Title: A Single-arm, Open-label, Multi-cohort, Multi-center Phase II Clinical Study of Anlotinib Combined With Penpulimab in the Treatment of Recurrent or Metastatic Gynecological Cancer
Brief Title: A Phase II Study of Anlotinib Combined With Penpulimab in Subjects With Gynecological Cancer
Acronym: ALTER-GO-020
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guonan Zhang, Director, Head of Gynecologic Oncology Center, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTERGO020
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Gynecological Cancer
MeSH Terms: interventions — penpulimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab+Anlotinib (Experimental): Penpulimab 200 mg IV on Day 1 of each 21-day cycle plus Anlotinib capsules 12mg given orally in fasting conditions , once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21)
  Interventions: Drug: Penpulimab; Drug: Anlotinib

INTERVENTIONS:
Drug: Penpulimab — Penpulimab is a humanized monoclonal antibody targeting programmed cell death-1 (PD-1), which prevents PD-1 from binding to PD-L1 and PD-L2 receptors on tumor cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Drug: Anlotinib — A multi-target receptor tyrosine kinase inhibitor

SUMMARY:
This is a single-arm, open-label, phase II clinical trial to evaluate the efficacy and safety of penpulimab combined with anlotinib in subjects with gynecological cancer, including 23 ovarian cancer，37 endometrial cancer，26 cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form;
* 18 years and older, female, Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1, life expectancy ≥3 months;
* Histopathologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal cancer; or endometrial cancer; or cervical cancer (including squamous cell, adenocarcinoma, or adenosquamous cell carcinoma);
* Patients must also meet any of the following conditions:

  1. Platinum-resistant relapsed or platinum-refractory ovarian cancer, the patient has received at least 1 line of platinum-based chemotherapy after previous cytoreductive surgery;
  2. With residual disease after surgery or inoperable stage III-IV endometrial cancer, and refused to receive chemoradiation/radiation/chemotherapy; or recurrent endometrial cancer unsuitable or refusing standard therapy;
  3. Persistent cervical cancer unsuitable for curative treatment, or recurrent/metastatic cervical cancer that refuses to receive standard treatment (for recurrent disease, not yet treated).
* At least one measurable lesion according to the RECIST 1.1;
* Try to provide tumor tissue samples for PD-L1 testing (not required)；
* Demonstrates adequate organ function:

  1. Blood routine inspection: Hemoglobin (HB) >= 90 g/L; The absolute value of neutrophil (ANC) >= 1.5x10^9/L;Platelets (PLT) >= 100x10^9/L;
  2. Blood biochemical inspection: Serum creatinine (Cr) <= 1.5 ULN, or creatinine clearance (CCr) >= 60mL / min; Total bilirubin (TBIL) <= 1.5 ULN, or direct bilirubin <= 1.0 ULN; AST and ALT <= 2.5 ULN.
  3. Blood coagulation function: Activated partial thromboplastin time, international standardized ratio adn prothrombin time <=1.5 ULN;
  4. Cardiac Function: left ventricular ejection fraction (LVEF) >=50%;
* Women of child-bearing potential must agree to use contraceptive measures (such as intrauterine devices or condoms) during the study and for 6 months after the end of the study, and have a negative serum pregnancy test within 7 days of enrollment, and must be non lactating subjects.

Exclusion Criteria:

* Has other non-epithelial ovarian tumors or borderline ovarian epithelial tumors; has carcinosarcoma, endometrial leiomyosarcoma, endometrial stromal sarcoma, or other high-grade sarcoma; has small cell carcinoma of the cervix, or clear cell carcinoma;
* Other malignant tumors that have appeared or are currently present within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors;
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137);
* Has received prior therapy with tyrosine kinase inhibitors that target VEGFR, such as pazopanib, sorafenib, regorafenib, apatinib and other drugs; but previous bevacizumab treatment is allowed (only for ovarian cancer cohorts), provided that the treatment is stopped for more than 4 weeks before enrollment;
* Has received prior radiotherapy within 4 weeks prior to enrollment (participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis - a 2-week washout is permitted for palliative radiation to non-CNS disease and vaginal brachytherapy);
* Has received prior hormonal therapy for the treatment of endometrial carcinoma within 1 week before enrollment;
* Expect to use any active vaccine against infectious diseases (such as influenza vaccine, chickenpox vaccine, etc.) within 28 days before the first dose or during the study period;
* Patients received systemic glucocorticoid therapy or other immunosuppressive therapy (dose> 10mg / day prednisone or other effective hormones) within 14 days before the first dose;
* Active autoimmune diseases that require systemic treatment have occurred within 2 years before the first dose;
* Subjects known to be allergic to the study drug or any of its excipients or have experienced a severe allergic reaction to other monoclonal antibodies;
* Has uncontrollable symptoms of brain metastases, spinal cord compression, cancerous meningitis;
* Has any bleeding or bleeding event ≥ CTC AE Grade 3 or unhealed wounds, ulcers or fractures within 4 weeks before enrollment;
* Patients with a clear tendency to gastrointestinal bleeding；
* Suspected or definite presence of symptoms or signs of radiation enteritis, and recurrence within 1 year from the end of radiotherapy;
* Patients whose tumors have invaded large blood vessels or poorly demarcated from the blood vessels according to imaging findings (CT/MRI);
* Prophylactic use of low dose aspirin (≤100mg/d) and low molecular weight heparin (≤40mg/d) is permitted in patients undergoing thrombolysis or anticoagulant therapy;
* Has clinically significant thyroid dysfunction before enrollment;
* Has multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
* Has any severe acute complications before enrollment:

  1. Blood pressure control is not ideal (systolic pressure >= 150 mmHg, diastolic pressure >= 100 mmHg);
  2. Patients had Unstable angina pectoris, myocardial infarction, ≥grade 2 congestive heart failure, or arrhythmia requiring treatment (including QTc ≥480 ms) within 6 months before enrollment;
  3. Active or uncontrolled serious infection (≥CTC AE grade 2 infection);
  4. Epidemiological test results during the screening period showed that any of the following is met: * HBsAg positive and HBV DNA exceeds the upper limit of normal value (those who fall within the normal range after antiviral treatment can be included); * Anti-HCV positive and HCV RNA positive; * HIV positive;
  5. Poorly controlled diabetes (fasting blood glucose ≥ grade 2);
  6. Had an arterio / venous thrombotic / carcinothrombotic event within 6 months, such as cerebrovascular accident (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, pulmonary embolism, and Hypertensive crisis or hypertensive encephalopathy;
  7. Exacerbated chronic obstructive pulmonary disease (COPD) or other respiratory diseases that require hospitalization, or have active lung infections and/or acute bacterial or fungal infections that require intravenous antibiotic treatment within 28 days before the first dose.
* Has participated in other anti-tumor intervention clinical trials within 4 weeks before the first medication;
* According to the judgement of the researchers, there are other factors that may lead to the termination of the study. For example, other serious diseases including mental disorders need to be treated together, serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR)

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 96 weeks
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.
Duration of Response (DOR) | up to 96 weeks
  Time from tumor first assessment to CR or PR to first assessment to PD (Progressive Disease) or death from any cause
Disease control rate（DCR） | up to 96 weeks
  Percentage of Participants Achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Overall Survival (OS) | up to 120 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Guonan Zhang, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangdong, Guangdong
  - The First Affiliated Hospital of USTC, Anhui Provincial Hospital, Hefei, Hefei
  - Shaanxi Provincial Cancer Hospital, Xi’an, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Sicchuan cancer hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No